CLINICAL TRIAL: NCT00800410
Title: A Pilot Randomized Diabetes Intervention Among Inner-city African American and Latino Adults
Brief Title: REACH Detroit Partnership Family Intervention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Michael Spencer, Associate Professor, University of Michigan School of Social Work
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: F012089-049555; 5P60DK020572 (NIH)
Record Dates: First submitted 2008-11-18; First posted 2008-12-02 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes Mellitus
Keywords: Randomized Controlled Trial
MeSH Terms: conditions — Diabetes Mellitus | interventions — Community Health Workers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Information on community resources (No Intervention): Participants received information about free and publicly available community resources on healthy lifestyle activities
- Community Health Worker services (Experimental)
  Interventions: Behavioral: Community Health Worker (CHW) services

INTERVENTIONS:
Behavioral: Community Health Worker (CHW) services — CHW services included access to an 11 week healthy lifestyle education curriculum, two home visits per month, two additional phone contacts per month, and accompanied participants to one clinic visit within the six month intervention period
  Arms: Community Health Worker services

SUMMARY:
The objectives of the proposed study are to determine whether culturally diverse community residents with diabetes are willing to participate in our community health worker intervention using randomized controlled trial (RCT) methods and to explore and document effective processes and protocols for RCT methods in these communities. The investigators will examine retention rates, identify reasons for attrition through interviews and focus groups, and determine strategies for improving recruitment, retention, and intervention methods. As a secondary objective, the investigators will explore the potential impacts of the intervention for improving healthy lifestyles, diabetes self-management, and selected health outcomes of participants.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Had physician-diagnosed type 2 diabetes
* Self-identified as African American or Latino/Hispanic
* Lived in the targeted zip codes.

Exclusion Criteria:

* Individuals who already had serious diabetes-related complications, such as blindness, amputated limbs, and kidney failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2004-09; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | 6 months

SECONDARY OUTCOMES:
LDL cholesterol | 6 months
Blood pressure | 6 months
Diabetes self-management knowledge | 6 months
Diabetes Self Management and Self Care Activities (physical activity, healthy eating, glucose testing, medication taking, required screening tests/exams) | 6 months
Diabetes specific emotional distress | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Spencer, PhD, MSW, Principal Investigator — University of Michigan
Locations (1):
- Community Health and Social Services (CHASS), Detroit, Michigan, United States

REFERENCES:
- [Derived] Spencer MS, Kieffer EC, Sinco B, Piatt G, Palmisano G, Hawkins J, Lebron A, Espitia N, Tang T, Funnell M, Heisler M. Outcomes at 18 Months From a Community Health Worker and Peer Leader Diabetes Self-Management Program for Latino Adults. Diabetes Care. 2018 Jul;41(7):1414-1422. doi: 10.2337/dc17-0978. Epub 2018 Apr 27. PMID 29703724
- [Derived] Rosland AM, Kieffer E, Spencer M, Sinco B, Palmisano G, Valerio M, Nicklett E, Heisler M. Do pre-existing diabetes social support or depressive symptoms influence the effectiveness of a diabetes management intervention? Patient Educ Couns. 2015 Nov;98(11):1402-9. doi: 10.1016/j.pec.2015.05.019. Epub 2015 Jun 5. PMID 26234800